CLINICAL TRIAL: NCT02250508
Title: A Randomised, Comparative, Single Dose, Open Study to Compare the Pharmacokinetics and Safety of Optivate® and Haemate P® in Patients With Different Types of Von Willebrand Disease.
Brief Title: A Study to Compare the Pharmacokinetics and Safety of Optivate® and Haemate P® in Patients With Von Willebrand Disease.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bio Products Laboratory (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 8VWF04
Record Dates: First submitted 2014-09-02; First posted 2014-09-26 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: vonWillebrand's Disease
MeSH Terms: interventions — optivate; Factor VIII; factor VIII, von Willebrand factor drug combination

ARMS (2):
- Optivate® (Experimental)
  Interventions: Biological: Optivate® (Human Coagulation Factor VIII)
- Haemate P® (Active Comparator)
  Interventions: Biological: Haemate P® (Human Coagulation Factor VIII)

INTERVENTIONS:
Biological: Optivate® (Human Coagulation Factor VIII)
  Arms: Optivate®
Biological: Haemate P® (Human Coagulation Factor VIII)
  Arms: Haemate P®

SUMMARY:
The main objectives of the study were

* to compare the pharmacokinetics (PK) of Optivate® and Haemate P® in various types of vonWillebrand disease (VWD) using the results from the VWF: RCo, VWF:Ag, VWF:CBA and Factor VIII assays.
* to compare the clinical tolerance and safety of these two treatments after single IV infusions in subjects with VWD.

ELIGIBILITY:
Inclusion Criteria:

* Previously treated subjects of at least 12 years of age, with any type of VWD were eligible for entry into this study.

Exclusion Criteria:

-

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-12; Primary Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
AUC (0-48h) for VWF: RCo | Pre-dose, 30 min, 1, 2, 5, 8, 24, 48 hours post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Hematology Dept., Sackler School of Medicine, Tel Aviv University, Tel Aviv, Israel

REFERENCES:
- See also: Related Info — http://www.bpl.co.uk